CLINICAL TRIAL: NCT02377739
Title: Non-invasive Ventilation in Patients With Interstitial Lung Disease - a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Weinmann Geräte für Medizin GmbH + Co. KG (Industry)
Responsible Party: Principal Investigator, Klaus Kenn, Dr. med. Klaus Kenn, Schön Klinik Berchtesgadener Land
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIV-ILD
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Noninvasive Ventilation; Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- non-invasive ventilation (Experimental): patients will undergo about 14 nights of non-invasive ventilation during pulmonary rehabilitation
  Interventions: Other: non-invasive ventilation

INTERVENTIONS:
Other: non-invasive ventilation — patients will undergo a nocturnal non-invasive ventilation

SUMMARY:
The efficiency of non-invasive ventilation (NIV) in hypercapnic patients with chronic obstructive pulmonary disease during pulmonary rehabilitation has been shown in numerous studies. There is only a limited number of therapeutic options for patients with severely progressed interstitial lung disease (ILD). The question whether chronic hypercapnic ILD-patients are able to profit from nocturnal NIV and thus increase their performance in physical training has been left unknown. Therefore, this study aims to evaluate the feasibility of the initialization of a NIV for hypercapnic ILD-patients during pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Interstitial lung disease
* Hypercapnia defined as carbon dioxide partial pressure ≥45 mmHg (at rest, night or activity)
* already existing but not sufficient and regular use of non-invasive ventilation (≤3h/24h)
* patients consent to participate in this trial

Exclusion Criteria:

* acute pulmonary insufficiency (ph<7.35)
* acute, clinically relevant heart disease
* already existing and sufficient use of non-invasive ventilation (≥3h/24h)
* Body-Mass-Index>30
* obstructive sleep apnea
* Intolerance to perform non-invasive ventilation
* acute infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
timespan until sufficient use of noninvasive ventilation > 6h during night | day 4-16

SECONDARY OUTCOMES:
6-minute walking test | day 1-3 and day 17-19
  change in 6-minute walking distance
arterial pressure of carbon dioxide during night | day 1-3 and day 17-19
  measured transcutaneously by a Sentec device
lung function measured by bodyplethysmograph | day 1-3 and 17-19
  measured by bodyplethysmograph
energy expenditure during night assessed by Sensewear Armband | day 5 and 15
  assessed by Sensewear Armband
quality of life | day 1-3 and 17-19
  Short-Form-36 health survey, Hospital Anxiety and Depression scale and severe respiratory insufficiency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, MD, Principal Investigator — Schoen Klinik Berchtesgadener Land
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany